CLINICAL TRIAL: NCT03106116
Title: A Prospective, Randomized Study of Enhanced External Counterpulsation Therapy on Ventricular Function in Patients With Coronary Heart Disease
Brief Title: Efficacy of Enhanced External Counterpulsation on Ventricular Function
Acronym: EECPVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yan Zhang, Associate professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EECP-3
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Heart Disease; Ventricular Function; Vascular Endothelium; Counterpulsation, External
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced External Counterpulsation (Experimental): Experimental: Enhanced External Counterpulsation (EECP) intervention on top of guideline- driven standard medical therapy for coronary heart disease
  Interventions: Device: Experimental: Enhanced External Counterpulsation; Drug: Standard medical therapy
- Control (Active Comparator): Guideline- driven standard medical therapy for 7 weeks without Enhanced External Counterpulsation intervention
  Interventions: Drug: Standard medical therapy

INTERVENTIONS:
Device: Experimental: Enhanced External Counterpulsation — Enhanced External Counterpulsation (EECP) is a technique for assisting the circulation by decreasing the afterload of the left ventricle and augmenting the diastolic pressure externally by applying a negative pressure to the lower extremities during cardiac systole. EECP therapy has been approved by the United States Food and Drug Administration (FDA) for the treatment of refractory angina and heart failure. Administration of 35-36 hours EECP therapy over a 7 week period, one hour session every working day.
  Other Names: EECP
  Arms: Enhanced External Counterpulsation
Drug: Standard medical therapy — Guideline- driven standard medical treatment for 7 weeks
  Other Names: Guideline- driven standard medical therapy

SUMMARY:
The purpose of this study is to investigate the efficacy of Enhanced External Counterpulsation (EECP) therapy on ventricular function in patients with coronary heart disease

DETAILED DESCRIPTION:
Patients with coronary heart disease will be randomized into two groups:

standard medical treatment and standard medical treatment plus EECP intervention. Ventricular structure and function will be measured and compared.

ELIGIBILITY:
Inclusion Criteria:

* More than 50% stenosis of left main trunk and 3 epicardial coronary arteries and their large branches showed by coronary angiography
* Or history of myocardial infarction
* Or history of prior revascularization
* Signed informed consent to participate in the study

Exclusion Criteria:

* Clinically significant valvular heart disease
* Aortic aneurysm
* Congenital heart disease
* Acute myocarditis
* Arrhythmias significantly interfere with the triggering of the EECP device
* History of cerebral hemorrhage
* Hemorrhagic disease
* Lower limb infection, phlebitis
* Deep venous thrombosis
* Malignant disease
* International normalized ratio (INR) > 2.5
* Uncontrolled hypertension, defined as systolic blood pressure > 180mmHg or diastolic blood pressure > 110mmHg
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Change in heart function | 7 weeks
  Change from baseline in heart function assessed by trans- thoracic echocardiography at 7 weeks

SECONDARY OUTCOMES:
Change in cardiac chamber diameter | 7 weeks
  Change from baseline in cardiac chamber diameterat 7 weeks
Change in ventricular wall thickness | 7 weeks
  Change from baseline in ventricular wall thickness

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, M. D., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Zhensheng Zheng, M. D., Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat- sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No